CLINICAL TRIAL: NCT01731600
Title: A Multinational, Open-Label, Non-Controlled Trial on Safety, Efficacy and Pharmacokinetics of NNC 0129-0000-1003 in Previously Treated Paediatric Patients With Severe Haemophilia A
Acronym: pathfinder™5
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN7088-3885; U1111-1129-6009 (Other: WHO); 2012-001711-23 (EudraCT Number); JapicCTI-132214 (Registry Identifier: JAPIC)
Record Dates: First submitted 2012-11-09; First posted 2012-11-22 (Estimated); Results first posted 2019-10-30 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- N8-GP (Experimental)
  Interventions: Drug: turoctocog alfa pegol

INTERVENTIONS:
Drug: turoctocog alfa pegol — Fixed dose of turoctocog alfa pegol for intravenous injections (i.v.) twice weekly for prophylaxis. In addition, turoctocog alfa pegol will be administered to treat bleeding episodes during the trial period. Bleeding episodes will be treated with doses of 20-75 U/kg body weight.
  Other Names: NNC 0129-0000-1003; N8-GP

SUMMARY:
This trial is conducted globally. The aim of the trial is to investigate safety, efficacy and pharmacokinetics (the exposure of the trial drug in the body) of NNC 0129-0000-1003 (N8-GP) in children with severe haemophilia A who have undergone treatment with previous factor VIII (FVIII) products.

ELIGIBILITY:
Inclusion Criteria:

* Male patients with severe congenital haemophilia A (FVIII activity level below 1%)
* Weight above or equal to 10 kg - Documented history of 150 exposure days (ED) to FVIII products for patients aged 6-11 years and above 50 ED to FVIII products for patients aged 0-5 years

Exclusion Criteria:

- Any history of FVIII inhibitors

Ages: 0 Years to 11 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2013-02-20 (Actual); Primary Completion 2014-09-15 (Actual); Study Completion 2018-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (50):
- United States (23):
  - Novo Nordisk Investigational Site, Phoenix, Arizona
  - Novo Nordisk Investigational Site, Long Beach, California
  - Novo Nordisk Investigational Site, Orange, California
  - Novo Nordisk Investigational Site, Washington D.C., District of Columbia
  - Novo Nordisk Investigational Site, Orlando, Florida
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, Boise, Idaho
  - Novo Nordisk Investigational Site, Iowa City, Iowa
  - Novo Nordisk Investigational Site, New Orleans, Louisiana
  - Novo Nordisk Investigational Site, Boston, Massachusetts
  - Novo Nordisk Investigational Site, Minneapolis, Minnesota
  - Novo Nordisk Investigational Site, Omaha, Nebraska
  - Novo Nordisk Investigational Site, New Hyde Park, New York
  - Novo Nordisk Investigational Site, Charlotte, North Carolina
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Dayton, Ohio
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Charleston, South Carolina
  - Novo Nordisk Investigational Site, Nashville, Tennessee
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Charlottesville, Virginia
  - Novo Nordisk Investigational Site, Spokane, Washington
- Novo Nordisk Investigational Site, Rio de Janeiro, Brazil
- Novo Nordisk Investigational Site, Toronto, Ontario, Canada
- France (3):
  - Novo Nordisk Investigational Site, Bron
  - Novo Nordisk Investigational Site, Lille
  - Novo Nordisk Investigational Site, Paris
- Greece (2):
  - Novo Nordisk Investigational Site, Athens
  - Novo Nordisk Investigational Site, Thessaloniki
- Novo Nordisk Investigational Site, Tel Litwinsky, Israel
- Novo Nordisk Investigational Site, Vicenza, Italy
- Japan (2):
  - Novo Nordisk Investigational Site, Kitakyusyu, Fukuoka
  - Novo Nordisk Investigational Site, Tokyo
- Novo Nordisk Investigational Site, Vilnius, Lithuania
- Novo Nordisk Investigational Site, Kuala Lumpur, Malaysia
- Novo Nordisk Investigational Site, Porto, Portugal
- Novo Nordisk Investigational Site, San Juan, Puerto Rico
- Switzerland (3):
  - Novo Nordisk Investigational Site, Bellinzona
  - Novo Nordisk Investigational Site, Lucerne
  - Novo Nordisk Investigational Site, Zurich
- Turkey (Türkiye) (4):
  - Novo Nordisk Investigational Site, Antalya
  - Novo Nordisk Investigational Site, Bornova-IZMIR
  - Novo Nordisk Investigational Site, İzmit
  - Novo Nordisk Investigational Site, Samsun
- Ukraine (2):
  - Novo Nordisk Investigational Site, Donetsk
  - Novo Nordisk Investigational Site, Lviv
- United Kingdom (3):
  - Novo Nordisk Investigational Site, Leicester
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Oxford

REFERENCES:
- [Result] Tosetto A, Neff A, Lentz SR, Santagostino E, Nemes L, Sathar J, Meijer K, Chowdary P, Shen C, Landorph A, Hampton K. Turoctocog alfa pegol provides effective management for major and minor surgical procedures in patients across all age groups with severe haemophilia A: Full data set from the pathfinder 3 and 5 phase III trials. Haemophilia. 2020 May;26(3):450-458. doi: 10.1111/hae.13980. Epub 2020 Apr 15. PMID 32293786
- [Result] Saulyte Trakymiene S, Economou M, Kenet G, Landorph A, Shen C, Kearney S. Long-term safety and efficacy of N8-GP in previously treated pediatric patients with hemophilia A: Final results from pathfinder5. J Thromb Haemost. 2020 Sep;18 Suppl 1(Suppl 1):15-25. doi: 10.1111/jth.15036. PMID 32940955
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 36 sites in 15 countries as follows: Canada (1), France (2), Germany (1), Greece (2 sites screened/1 site randomised subjects), Israel (1), Italy (1), Japan (2), Lithuania (1), Malaysia (1), Portugal (1), Switzerland (3), Turkey (3), Ukraine (2), United Kingdom (3), and United States (12).
Groups:
- Younger Children (0 - 5 Years): Participants (0 - 5 years) previously treated with FVIII received N8-GP (prophylaxis or treatment of bleeding episodes). Prophylaxis: N8-GP as a single bolus iv injection 60 IU/kg twice weekly. Treatment of bleeding episodes: N8-GP ranging from 20-75 IU/kg, according to severity and location of bleeding episode. The trial consisted of main and extension phase. Duration of main phase for each subject was approximately 26 weeks (50 exposure days). After completion of main phase, subjects could continue until the end of the extension phase, which was defined as LPLV. All subjects continued twice weekly or every third day prophylaxis regimen in extension phase as prescribed for main phase. However, after 12 months treatment with N8-GP (main phase+extension phase) the investigator was permitted to prescribe extra coverage before physical activities.
- Older Children (6 - 11 Years): Participants (6 - 11 years) previously treated with FVIII received N8-GP (prophylaxis or treatment of bleeding episodes). Prophylaxis: N8-GP as a single bolus iv injection 60 IU/kg twice weekly. Treatment of bleeding episodes: N8-GP ranging from 20-75 IU/kg, according to severity and location of bleeding episode. The trial consisted of main and extension phase. Duration of main phase for each subject was approximately 26 weeks (50 exposure days). After completion of main phase, subjects could continue until the end of the extension phase, which was defined as LPLV. All subjects continued twice weekly or every third day prophylaxis regimen in extension phase as prescribed for main phase. However, after 12 months treatment with N8-GP (main phase+extension phase) the investigator was permitted to prescribe extra coverage before physical activities.
Period: Overall Study
Arm/Group | Younger Children (0 - 5 Years) | Older Children (6 - 11 Years)
Started | 34 | 34
Completed | 28 | 34
Not Completed | 6 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal criteria | 1 | 0
Not completed — Other reasons | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Younger Children (0 - 5 Years) | Older Children (6 - 11 Years) | Total
Number analyzed (Participants) | 34 | 34 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.0 (1.3) | 8.9 (1.7) | 6.0 (3.3)
Age, Customized [Count of Participants; unit: Participants]
  Infants and toddlers (28 days-23 months) | 6 | 0 | 6
  Children (2-11 years) | 28 | 34 | 62
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 34 | 34 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 34 | 30 | 64
  Unknown or Not Reported | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race of the participants
  Participants
    White | 30 | 25 | 55
    Black or African American | 2 | 1 | 3
    Asian | 1 | 4 | 5
    Other | 1 | 1 | 2
    Not applicable | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Inhibitory Antibodies Against Coagulation Factor VIII (FVIII) ≥0.6 Bethesda Units
Description: The number of participants with inhibitory antibodies against coagulation factor VIII (FVIII) ≥0.6 Bethesda units was presented.
Time Frame: During the main phase of the trial (from 0-26 weeks of treatment)
Population: Results were based on safety analysis set (SAS). The SAS consists of all patients exposed to at least one dose of turoctocog alfa pegol. Number analysed = participants with minimum of 50 exposure days and developed inhibitory antibodies
Measure: Number; unit: Participants
Groups:
- Younger Children (0 - 5 Years) [Main Trial]: Participants (0 - 5 years) previously treated with FVIII received N8-GP (prophylaxis or treatment of bleeding episodes). The trial consisted of main and extension phase. Duration of main phase for each subject was approximately 26 weeks (50 exposure days).
- Older Children (6 - 11 Years) [Main Trial]: Participants (6 - 11 years) previously treated with FVIII received N8-GP (prophylaxis or treatment of bleeding episodes). The trial consisted of main and extension phase. Duration of main phase for each subject was approximately 26 weeks (50 exposure days).
Arm/Group | Younger Children (0 - 5 Years) [Main Trial] | Older Children (6 - 11 Years) [Main Trial]
Number analyzed (Participants) | 34 | 34
Participants | 0 | 0
Statistical Analysis 1: Comparison: Younger Children (0 - 5 Years) [Main Trial] vs Older Children (6 - 11 Years) [Main Trial]; A one-sided, upper 97.5% confidence limit was provided based on an exact calculation in the binomial distribution; Test type: Other; Incidence rate = 0, 97.5% CI 1-sided [upper limit 0.067] — The incidence of inhibitory antibodies was calculated as number of patients with inhibitors during the main phase of the trial divided by number of patients in the main phase of the trial

2. Secondary Outcome: Frequency of Adverse Events Including Serious Adverse Events Reported During the Trial Period
Description: The frequency of adverse events including serious adverse events reported during the main and extension phase of the trial. The data presented is the rate of AE i.e. number of AEs per patient years of exposue.
Time Frame: Main phase: (from 0-26 weeks of treatment) and full trial: (0 weeks to last patient's completion of the trial, an average of 4.5 years)
Population: Results were based on SAS.
Measure: Number; unit: Events per patient years of exposure
Groups:
- Younger Children (0 - 5 Years) [Full Trial]: Participants (0 - 5 years) previously treated with FVIII received N8-GP (prophylaxis or treatment of bleeding episodes). The trial consisted of main and extension phase. Duration of main phase for each subject was approximately 26 weeks (50 exposure days). After completion of main phase, subjects could continue until the end of the extension phase, which was defined as LPLV. All subjects continued twice weekly or every third day prophylaxis regimen in extension phase as prescribed for main phase. However, after 12 months treatment with N8-GP (main phase+extension phase) the investigator was permitted to prescribe extra coverage before physical activities.
- Older Children (6 - 11 Years) [Full Trial]: Participants (6 - 11 years) previously treated with FVIII received N8-GP (prophylaxis or treatment of bleeding episodes). The trial consisted of main and extension phase. Duration of main phase for each subject was approximately 26 weeks (50 exposure days). After completion of main phase, subjects could continue until the end of the extension phase, which was defined as LPLV. All subjects continued twice weekly or every third day prophylaxis regimen in extension phase as prescribed for main phase. However, after 12 months treatment with N8-GP (main phase+extension phase) the investigator was permitted to prescribe extra coverage before physical activities.
Arm/Group | Younger Children (0 - 5 Years) [Main Trial] | Older Children (6 - 11 Years) [Main Trial] | Younger Children (0 - 5 Years) [Full Trial] | Older Children (6 - 11 Years) [Full Trial]
Number analyzed (Participants) | 34 | 34 | 34 | 34
Events per patient years of exposure | 4.87 | 4.74 | 3.09 | 2.45

3. Secondary Outcome: Haemostatic Effect of N8-GP When Used for Treatment of Bleeding Episodes and Assessed as: Excellent, Good, Moderate, or None
Description: Haemostatic effect of N8-GP for treatment of bleeding episodes was assessed by 4-point response scale: none, moderate, good or excellent. Evaluation during trial was done by patient and/or parent(s)/caregiver 8 hours after first injection as follows: Excellent: Abrupt pain relief and/or clear improvement in objective signs of bleeding within approximately 8 hours after a single injection; Good: Definite pain relief and/or improvement in signs of bleeding within approximately 8 hours after a single injection, but possibly requiring more than one injection for complete resolution; Moderate: Probable or slight beneficial effect within approximately 8 hours after the first injection, but usually requiring more than one injection; None: No improvement, or worsening of symptoms.
Time Frame: as for outcome 2
Population: Results were based on full analysis set (FAS). All trial patients allocated to treatment, for which at least one of the pharmacokinetic or efficacy endpoints was assessed, were included in the FAS.
Measure: Count of Units; unit: Bleeding episodes
Units Other Than Participants: Bleeding episodes
Arm/Group | Younger Children (0 - 5 Years) [Main Trial] | Older Children (6 - 11 Years) [Main Trial] | Younger Children (0 - 5 Years) [Full Trial] | Older Children (6 - 11 Years) [Full Trial]
Number analyzed (Participants) | 34 | 34 | 34 | 34
Number analyzed (Bleeding episodes) | 30 | 40 | 108 | 222
Bleeding episodes
  Excellent | 11 | 12 | 47 | 96
  Good | 13 | 19 | 48 | 74
  Moderate | 4 | 7 | 9 | 44
  None | 1 | 0 | 2 | 2
  Missing | 1 | 2 | 2 | 6

4. Secondary Outcome: Number of Bleeding Episodes During Prophylactic Treatment With N8-GP (Annualised Bleeding Rate)
Description: The number of bleeding episodes per year reported during the prophylactic treatment with N8-GP.
Time Frame: as for outcome 2
Population: Results were based on FAS.
Measure: Median (Inter-Quartile Range); unit: bleeds/patient/year
Arm/Group | Younger Children (0 - 5 Years) [Main Trial] | Older Children (6 - 11 Years) [Main Trial] | Younger Children (0 - 5 Years) [Full Trial] | Older Children (6 - 11 Years) [Full Trial]
Number analyzed (Participants) | 34 | 34 | 34 | 34
bleeds/patient/year | 1.94 [0.00 to 2.08] | 1.97 [0.00 to 3.91] | 0.61 [0.20 to 1.19] | 0.93 [0.20 to 2.11]

5. Secondary Outcome: Consumption of N8-GP Per Bleeding Episode (Number of Injections)
Description: The mean number of injections of N8-GP used for treatment of a bleed from start to stop of a bleed.
Time Frame: as for outcome 2
Population: Results were based on FAS.
Measure: Mean (Standard Deviation); unit: Number of injections
Units Other Than Participants: Bleeding episodes
Arm/Group | Younger Children (0 - 5 Years) [Main Trial] | Older Children (6 - 11 Years) [Main Trial] | Younger Children (0 - 5 Years) [Full Trial] | Older Children (6 - 11 Years) [Full Trial]
Number analyzed (Participants) | 34 | 34 | 34 | 34
Number analyzed (Bleeding episodes) | 30 | 40 | 108 | 222
Number of injections | 1.9 (1.5) | 1.6 (0.9) | 1.6 (1.3) | 1.5 (1.1)

6. Secondary Outcome: Consumption of N8-GP Per Bleeding Episode (U/kg)
Description: The mean consumption of N8-GP used for treatment of a bleed from start to stop of a bleed.
Time Frame: as for outcome 2
Population: Results were based on FAS.
Measure: Mean (Standard Deviation); unit: IU/kg/bleed
Units Other Than Participants: Bleeding episodes
Arm/Group | Younger Children (0 - 5 Years) [Main Trial] | Older Children (6 - 11 Years) [Main Trial] | Younger Children (0 - 5 Years) [Full Trial] | Older Children (6 - 11 Years) [Full Trial]
Number analyzed (Participants) | 34 | 34 | 40 | 34
Number analyzed (Bleeding episodes) | 30 | 40 | 108 | 222
IU/kg/bleed | 123 (104.9) | 99 (54.4) | 102.8 (81) | 91 (58.3)

7. Secondary Outcome: Consumption of N8-GP During Prophylaxis (Number of Injections)
Description: The mean number of injections of N8-GP used for treatment of a bleed from start to stop of a bleed during prophylaxis.
Time Frame: as for outcome 2
Population: Results were based on FAS.
Measure: Mean (Standard Deviation); unit: Number of injections
Units Other Than Participants: Injections
Arm/Group | Younger Children (0 - 5 Years) [Main Trial] | Older Children (6 - 11 Years) [Main Trial] | Younger Children (0 - 5 Years) [Full Trial] | Older Children (6 - 11 Years) [Full Trial]
Number analyzed (Participants) | 34 | 34 | 34 | 34
Number analyzed (Injections) | 1592 | 1799 | 14442 | 17243
Number of injections | 65.3 (6.5) | 62.3 (7.4) | 65.4 (7.5) | 64.1 (5.3)

8. Secondary Outcome: Consumption of N8-GP During Prophylaxis (U/kg Per Month)
Description: The mean consumption of N8-GP used for treatment of a bleed from start to stop of a bleed during prophylaxis (per month per subject). Consumption used for treatment includes all doses given (prophylaxis, treatment of bleed, minor surgery and pharmacokinetics [PK])
Time Frame: as for outcome 2
Population: Results were based on FAS.
Measure: Mean (Standard Deviation); unit: U/kg/month
Arm/Group | Younger Children (0 - 5 Years) [Main Trial] | Older Children (6 - 11 Years) [Main Trial] | Younger Children (0 - 5 Years) [Full Trial] | Older Children (6 - 11 Years) [Full Trial]
Number analyzed (Participants) | 34 | 34 | 34 | 34
U/kg/month | 572.5 (97.4) | 555.8 (44.6) | 564.9 (86.6) | 563.4 (15.1)

9. Secondary Outcome: Consumption of N8-GP During Prophylaxis (U/kg Per Year)
Description: The mean consumption of N8-GP used for treatment of a bleed from start to stop of a bleed during prophylaxis (per year per subject). Consumption used for treatment includes all doses given (prophylaxis, treatment of bleed, minor surgery and pharmacokinetics)
Time Frame: as for outcome 2
Population: Results were based on FAS.
Measure: Mean (Standard Deviation); unit: U/kg/year
Arm/Group | Younger Children (0 - 5 Years) [Main Trial] | Older Children (6 - 11 Years) [Main Trial] | Younger Children (0 - 5 Years) [Full Trial] | Older Children (6 - 11 Years) [Full Trial]
Number analyzed (Participants) | 34 | 34 | 34 | 34
U/kg/year | 6870.3 (1169) | 6669.6 (535.8) | 6778.6 (1039) | 6760.4 (181.8)

10. Secondary Outcome: Incremental Recovery (Defined as the Peak Level Recorded 60 Min After End of Injection) Evaluated for Previous FVIII Product
Description: The incremental recovery was defined as the increase in plasma FVIII activity per IU/kg of factor administered recorded 60 minutes after end of injection. It was calculated as (Factor VIII procoagulant [FVIII:C] activity measured in plasma 60 min after dosing - FVIII:C activity measured in plasma immediately before dosing) / (dose injected at time 0 min), where the dose was expressed as U FVIII product per kg body weight. A chromogenic assay with normal human plasma (NHP) as calibrator was used.
Time Frame: 2-6 weeks prior to initial dosing with N8-GP and up to 30 hours after administration of previous FVIII product
Population: Results were based on FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: (IU/mL)/(U/kg)
Arm/Group | Younger Children (0 - 5 Years) [Full Trial] | Older Children (6 - 11 Years) [Full Trial]
Number analyzed (Participants) | 34 | 34
(IU/mL)/(U/kg) | 0.017 [0.014 to 0.021] | 0.022 [0.018 to 0.027]

11. Secondary Outcome: Incremental Recovery (Defined as the Peak Level Recorded 60 Min After End of Injection) Evaluated for N8-GP
Description: The incremental recovery was defined as the peak level recorded 60 min after end of injection and dose-normalised. It was calculated as (FVIII:C activity measured in plasma 60 min after dosing - FVIII:C activity measured in plasma immediately before dosing) / (dose injected at time 0 min), where the dose was expressed as U FVIII product per kg body weight. A chromogenic assay with product specific calibrator (PSS) as calibrator was used.
Time Frame: From 1 hour prior to and up to 96 hours after initial administration of N8-GP
Population: Results were based on FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: (IU/mL)/(U/kg)
Arm/Group | Younger Children (0 - 5 Years) [Full Trial] | Older Children (6 - 11 Years) [Full Trial]
Number analyzed (Participants) | 34 | 34
(IU/mL)/(U/kg) | 0.018 [0.015 to 0.022] | 0.020 [0.016 to 0.024]

12. Secondary Outcome: Area Under the Curve Evaluated for Previous FVIII Product
Description: Area under the curve (AUC) versus time from zero to infinity. This is calculated as AUC = AUClast + (C(t) / λz), where C(t) is the last measurable concentration. A chromogenic assay with NHP as calibrator was used.
Time Frame: 2-6 weeks prior to initial dosing with N8-GP and up to 30 hours after administration of previous FVIII product
Population: Results were based on FAS
Measure: Least Squares Mean (95% Confidence Interval); unit: IU×h/mL
Arm/Group | Younger Children (0 - 5 Years) [Full Trial] | Older Children (6 - 11 Years) [Full Trial]
Number analyzed (Participants) | 34 | 34
IU×h/mL | 11.628 [9.170 to 14.744] | 12.203 [9.336 to 15.951]

13. Secondary Outcome: Area Under the Curve Evaluated for N8-GP
Description: Area under the curve versus time from zero to infinity. This is calculated as AUC = AUClast + (C(t) / λz), where C(t) is the last measurable concentration. A chromogenic assay with product specific standard (PSS) as calibrator was used.
Time Frame: From 1 hour prior to and up to 96 hours after initial administration of N8-GP
Population: Results were based on FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: IU*h/mL
Arm/Group | Younger Children (0 - 5 Years) [Full Trial] | Older Children (6 - 11 Years) [Full Trial]
Number analyzed (Participants) | 34 | 34
IU*h/mL | 21.489 [16.785 to 27.511] | 25.026 [19.145 to 32.713]

14. Secondary Outcome: Terminal Half-life Evaluated for Previous FVIII Product
Description: t½ = ln(2) / λz, where t½ is terminal half-life and λz is the terminal elimination rate. The terminal elimination rate was planned estimated using linear regression on the terminal part of the time versus log(concentration) curve. A population-based method simultaneously estimating individual t½ values for all patients was applied, including patients with few values above the lower limit of quantification (LLOQ). This was estimated using time points from 1h to 30h. A chromogenic assay with PSS as calibrator was used.
Time Frame: 2-6 weeks prior to initial dosing with N8-GP and up to 30 hours after administration of previous FVIII product
Population: Results were based on FAS.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Younger Children (0 - 5 Years) [Full Trial] | Older Children (6 - 11 Years) [Full Trial]
Number analyzed (Participants) | 34 | 34
hours | 7.2 (20.1) | 7.5 (19.1)

15. Secondary Outcome: Terminal Half-life Evaluated for N8-GP
Description: t½ = ln(2) / λz, where λz is the terminal elimination rate. The terminal elimination rate was planned estimated using linear regression on the terminal part of the time versus log(concentration) curve. A population-based method simultaneously estimating individual t½ values for all patients was applied, including patients with few values above the LLOQ. This was estimated using time points from 6h to 96h. A chromogenic assay with PSS as calibrator was used.
Time Frame: From 1 hour prior to and up to 96 hours after initial administration of N8-GP
Population: Results were based on FAS.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Younger Children (0 - 5 Years) [Full Trial] | Older Children (6 - 11 Years) [Full Trial]
Number analyzed (Participants) | 34 | 34
hours | 13.6 (20.4) | 14.1 (25.0)

16. Secondary Outcome: Clearance Evaluated for Previous FVIII Product
Description: Total plasma clearance of drug after intravenous administration measured as actual dose/AUC. A chromogenic assay with NHP as calibrator was used.
Time Frame: 2-6 weeks prior to initial dosing with N8-GP and up to 30 hours after administration of previous FVIII product
Population: Results were based on FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/h/kg
Arm/Group | Younger Children (0 - 5 Years) [Full Trial] | Older Children (6 - 11 Years) [Full Trial]
Number analyzed (Participants) | 34 | 34
mL/h/kg | 4.322 [3.404 to 5.486] | 3.867 [2.955 to 5.061]

17. Secondary Outcome: Clearance Evaluated for N8-GP
Description: Total plasma clearance of drug after intravenous administration measured as actual dose/AUC. A chromogenic assay with PSS as calibrator was used.
Time Frame: From 1 hour prior to and up to 96 hours after initial administration of N8-GP.
Population: Results were based on FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/h/kg
Arm/Group | Younger Children (0 - 5 Years) [Full Trial] | Older Children (6 - 11 Years) [Full Trial]
Number analyzed (Participants) | 34 | 34
mL/h/kg | 2.601 [2.030 to 3.333] | 2.386 [1.823 to 3.123]

ADVERSE EVENTS:
Time Frame: From first exposure to N8-GP (visit 2) of main phase to end of extension phase (>=4 days after last dose of N8-GP, up to 4.5 years).
Description: The safety analysis set consists of all patients exposed to at least one dose of N8-GP.
Arm/Group | Younger Children£(0-5 Years) | Older Children£(6-11 Years)
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/34
Serious Adverse Events (participants affected / at risk) | 11/34 | 5/34
Other Adverse Events (participants affected / at risk) | 33/34 | 33/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Younger Children£(0-5 Years) (N=34) | Older Children£(6-11 Years) (N=34)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acquired phimosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (2) | 0 (0)
Encephalitis (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Sepsis syndrome (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Younger Children£(0-5 Years) (N=34) | Older Children£(6-11 Years) (N=34)
Abdominal pain (Gastrointestinal disorders) | 5 (7) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (5)
Acute sinusitis (Infections and infestations) | 0 (0) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 4 (5)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (2) | 2 (2)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (3) | 3 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 1 (1)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 3 (3) | 1 (1)
Bronchitis (Infections and infestations) | 3 (5) | 3 (3)
Cerumen impaction (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Chapped lips (Gastrointestinal disorders) | 0 (0) | 2 (2)
Conjunctivitis (Infections and infestations) | 2 (2) | 2 (2)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 3 (4)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (5)
Contusion (Injury, poisoning and procedural complications) | 4 (4) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (26) | 6 (6)
Dental caries (Gastrointestinal disorders) | 3 (5) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 5 (7) | 4 (5)
Ear infection (Infections and infestations) | 5 (5) | 3 (5)
Ear pain (Ear and labyrinth disorders) | 4 (5) | 1 (2)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (28) | 1 (3)
Erythema (Skin and subcutaneous tissue disorders) | 3 (5) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (3)
Fall (Injury, poisoning and procedural complications) | 5 (8) | 3 (4)
Food allergy (Immune system disorders) | 1 (2) | 2 (4)
Gastroenteritis (Infections and infestations) | 7 (10) | 9 (13)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 2 (2)
Haematoma (Vascular disorders) | 2 (2) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 3 (4) | 4 (5)
Headache (Nervous system disorders) | 5 (6) | 9 (16)
Hyperthermia (General disorders) | 2 (2) | 1 (1)
Influenza (Infections and infestations) | 5 (9) | 6 (10)
Joint injury (Injury, poisoning and procedural complications) | 2 (2) | 3 (4)
Joint swelling (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 5 (6)
Limb injury (Injury, poisoning and procedural complications) | 5 (5) | 4 (12)
Molluscum contagiosum (Infections and infestations) | 2 (2) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2)
Nasopharyngitis (Infections and infestations) | 11 (21) | 10 (16)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 8 (10)
Otitis media (Infections and infestations) | 4 (4) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (11) | 6 (8)
Penile adhesion (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 3 (3)
Pharyngitis (Infections and infestations) | 2 (2) | 1 (2)
Pharyngitis streptococcal (Infections and infestations) | 2 (2) | 1 (2)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 7 (16) | 6 (9)
Rash (Skin and subcutaneous tissue disorders) | 7 (11) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rhinitis (Infections and infestations) | 8 (8) | 4 (7)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (4)
Seasonal allergy (Immune system disorders) | 2 (2) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1) | 2 (2)
Skin abrasion (Injury, poisoning and procedural complications) | 2 (2) | 3 (4)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Tonsillitis (Infections and infestations) | 2 (2) | 2 (5)
Upper respiratory tract infection (Infections and infestations) | 10 (20) | 13 (31)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Varicella (Infections and infestations) | 6 (6) | 1 (1)
Viral infection (Infections and infestations) | 4 (5) | 3 (3)
Viral pharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 4 (5) | 3 (5)
Vomiting (Gastrointestinal disorders) | 9 (10) | 3 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property

DOCUMENTS (1):
  • Study Protocol (2015-11-13): https://cdn.clinicaltrials.gov/large-docs/00/NCT01731600/Prot_000.pdf